CLINICAL TRIAL: NCT01373281
Title: Efficacy and Safety of a Novel Tetravalent Dengue Vaccine in Healthy Children Aged 2 to 14 Years in Asia
Brief Title: Study of a Novel Tetravalent Dengue Vaccine in Healthy Children Aged 2 to 14 Years in Asia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD14; UTN: U1111-1116-4957 (Other: WHO); 2014-001708-24 (EudraCT Number)
Record Dates: First submitted 2011-06-08; First posted 2011-06-14 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue; Dengue fever; Dengue Hemorrhagic Fever; CYD dengue vaccine; Flavivirus
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dengue Vaccine Group (Experimental): Participants were to receive CYD dengue vaccine at 0, 6, and 12 months.
  Interventions: Biological: Live, attenuated, dengue serotype 1, 2, 3, 4 virus
- Control Group (Placebo Comparator): Participants were to receive a placebo vaccine at 0, 6, and 12 months.
  Interventions: Biological: Placebo: Sodium chloride (NaCl) 0.9%

INTERVENTIONS:
Biological: Live, attenuated, dengue serotype 1, 2, 3, 4 virus — 0.5 mL, Subcutaneous
  Other Names: CYD Dengue Vaccine
  Arms: Dengue Vaccine Group
Biological: Placebo: Sodium chloride (NaCl) 0.9% — 0.5 mL, Subcutaneous
  Arms: Control Group

SUMMARY:
The aim of the trial was to assess the efficacy of the CYD dengue vaccine in preventing symptomatic, virologically-confirmed dengue (VCD) cases.

Primary Objective:

To assess the efficacy of CYD dengue vaccine after 3 vaccinations at 0, 6, and 12 months in preventing symptomatic VCD cases, regardless of the severity, due to any of the four serotypes in children aged 2 to 14 years at the time of inclusion.

Secondary Objectives:

* To describe the efficacy of CYD dengue vaccine in preventing symptomatic VCD cases after the third dose to the end of the Active Phase, after at least 1 dose, and after 2 doses.
* To describe the occurrence of serious adverse events (SAEs), including SAEs of special interest in all participants throughout the trial period.
* To describe the occurrence of hospitalized virologically-confirmed dengue (VCD) cases and the occurrence of severe (clinically-severe or as per World Health Organization (WHO) criteria) VCD cases, throughout the Surveillance Expansion period (SEP) and throughout the trial (from Day 0 to the end of the study).
* To describe the antibody response to each dengue serotype after Dose 2, after Dose 3, and 1 and 5 years after Dose 3.

DETAILED DESCRIPTION:
Participants were randomized to either receive 3 injections of CYD dengue vaccine or a placebo at 0, 6, and 12 months.

A subset of participants from each country were also evaluated for reactogenicity and immunogenicity.

Participants who consented to participate in the SEP were actively followed for dengue case detection (i.e. at least weekly contact and capturing any acute febrile illness, not just hospitalized febrile cases, as in the Active Phase). The SEP was designed to maximize the detection of symptomatic confirmed dengue (hospitalized or not) in order to describe CYD dengue vaccine efficacy and safety in preventing symptomatic dengue. Participants who declined participating in the SEP continued surveillance as in the Hospital Phase until trial completion.

Symptomatic VCD cases occurring more than (>) 28 days after dose 3 (during the Active Phase) are defined as:

* Acute febrile illness (i.e. temperature >=38 C on at least 2 consecutive days)
* Virologically confirmed by dengue Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) and/or dengue non-structural (NS)1 enzyme-linked immunosorbent assay (ELISA) Ag test

  1997 WHO Classification Dengue hemorrhagic fever (DHF) cases were defined as per the 1997 WHO criteria of clinical manifestations; a) Fever: acute onset, high (>= 38°C) and continuous, lasting 2 to 7 days and (b) any of the pre-listed hemorrhagic manifestations and laboratory findings of thrombocytopenia (platelet<=100 x 109/L) and plasma leakage as shown by hemoconcentation (hematocrit increased by 20 percent [%] or more) or pleural effusion (seen on chest X-ray [CXR]) and/or ascites and/or hypoaluminemia. The first two clinical criteria plus thrombocytopenia and signs of plasma leakage are enough to establish a clinical diagnosis of DHF.

DHF was graded as follows:- Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test; Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participants, usually in the form of skin and/or other hemorrhages; Grade III: Circulatory failure manifested by rapid and weak pulse, narrowing of pulse pressure (20 mmHg or less) or hypotension, with the presence of cold clammy skin and restlessness; and Grade IV: Profound shock with undetectable blood pressure and pulse.

Independent Data Monitoring Committee (IDMC) severity criteria The severity of VCD cases was assessed by an Independent IDMC using pre-defined standardized criteria. Following manifestations of severity were considered in all suspected VCD cases; 1) Platelet count <= 100000μl and bleeding (tourniquet, petechiae or any bleeding) plus plasma leakage (effusion on CXR OR clinically apparent ascites or hematocrit >=20% above baseline recovery level) 2) Shock (pulse pressure <= 20 mmHg in a child, or hypotension [<= 90 mmHg] with tachycardia, weak pulse and poor perfusion) 3) Bleeding requiring blood transfusion 4) Encephalopathy i.e. Unconsciousness or poor conscious state or convulsionsfitting not attributable to simple febrile convulsion as defined in the guidelines for definition and collection of febrile convulsions or focal neurological signs. Poor conscious state or unconsciousness must be supported by Glasgow Coma Scale (GCS) score. 5) Liver impairment (aspartate aminotransferase [AST] >1000IU/L or prothrombin time [PT] International normalized ratio [INR] >1.5) excluding other causes of viral hepatitis 6) Impaired kidney function (serum creatinine ≥ 1.5 mg/dL) 7) Myocarditis, pericarditis or clinical heart failure supported by CXR, echocardiography, electrocardiogram (ECG) or cardiac enzymes.

The designation of such cases as severe or otherwise will be made on a case by case basis by the IDMC.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 14 years on the day of inclusion and resident of the site zone
* Participant was in good health, based on medical history and physical examination
* Assent form or informed consent form has been signed and dated by the participant (based on local regulations), and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations)
* Participant attended all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or was of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination)
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Self-reported or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV) infection
* Self-reported systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as a site employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member (i.e., immediate, husband, wife and their children, adopted or natural) of the site employees or the Investigator.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10275 (Actual)
Dates: Start 2011-06-03 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (12):
- Indonesia (3):
  - Denpasar, Bali
  - Bandung, West Java
  - Jakarta
- Malaysia (2):
  - Kuala Lumpur
  - Pulau Pinang
- Philippines (2):
  - Cebu City
  - San Pablo
- Thailand (3):
  - Nai Muang, Changwat Kamphaeng Phet
  - Ban Pong, Changwat Ratchaburi
  - Photharam, Changwat Ratchaburi
- Vietnam (2):
  - Long Xuyen, An Giang
  - Mỹ Tho, Tien Giang Province

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Capeding MR, Tran NH, Hadinegoro SR, Ismail HI, Chotpitayasunondh T, Chua MN, Luong CQ, Rusmil K, Wirawan DN, Nallusamy R, Pitisuttithum P, Thisyakorn U, Yoon IK, van der Vliet D, Langevin E, Laot T, Hutagalung Y, Frago C, Boaz M, Wartel TA, Tornieporth NG, Saville M, Bouckenooghe A; CYD14 Study Group. Clinical efficacy and safety of a novel tetravalent dengue vaccine in healthy children in Asia: a phase 3, randomised, observer-masked, placebo-controlled trial. Lancet. 2014 Oct 11;384(9951):1358-65. doi: 10.1016/S0140-6736(14)61060-6. Epub 2014 Jul 10. PMID 25018116
- [Result] L'Azou M, Moureau A, Sarti E, Nealon J, Zambrano B, Wartel TA, Villar L, Capeding MR, Ochiai RL; CYD14 Primary Study Group; CYD15 Primary Study Group. Symptomatic Dengue in Children in 10 Asian and Latin American Countries. N Engl J Med. 2016 Mar 24;374(12):1155-66. doi: 10.1056/NEJMoa1503877. PMID 27007959
- [Result] Coudeville L, Baurin N, Vergu E. Estimation of parameters related to vaccine efficacy and dengue transmission from two large phase III studies. Vaccine. 2016 Dec 7;34(50):6417-6425. doi: 10.1016/j.vaccine.2015.11.023. Epub 2015 Nov 21. PMID 26614588
- [Result] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- [Result] Guy B, Jackson N. Dengue vaccine: hypotheses to understand CYD-TDV-induced protection. Nat Rev Microbiol. 2016 Jan;14(1):45-54. doi: 10.1038/nrmicro.2015.2. Epub 2015 Dec 7. PMID 26639777
- [Result] Gailhardou S, Skipetrova A, Dayan GH, Jezorwski J, Saville M, Van der Vliet D, Wartel TA. Safety Overview of a Recombinant Live-Attenuated Tetravalent Dengue Vaccine: Pooled Analysis of Data from 18 Clinical Trials. PLoS Negl Trop Dis. 2016 Jul 14;10(7):e0004821. doi: 10.1371/journal.pntd.0004821. eCollection 2016 Jul. PMID 27414655
- [Result] Vigne C, Dupuy M, Richetin A, Guy B, Jackson N, Bonaparte M, Hu B, Saville M, Chansinghakul D, Noriega F, Plennevaux E. Integrated immunogenicity analysis of a tetravalent dengue vaccine up to 4 y after vaccination. Hum Vaccin Immunother. 2017 Sep 2;13(9):2004-2016. doi: 10.1080/21645515.2017.1333211. Epub 2017 Jun 9. PMID 28598256
- [Result] Guy B, Noriega F, Ochiai RL, L'azou M, Delore V, Skipetrova A, Verdier F, Coudeville L, Savarino S, Jackson N. A recombinant live attenuated tetravalent vaccine for the prevention of dengue. Expert Rev Vaccines. 2017 Jul;16(7):1-13. doi: 10.1080/14760584.2017.1335201. Epub 2017 Jun 7. PMID 28590795
- [Result] Nealon J, Taurel AF, Capeding MR, Tran NH, Hadinegoro SR, Chotpitayasunondh T, Chong CK, Wartel TA, Beucher S, Frago C, Moureau A, Simmerman M, Laot T, L'Azou M, Bouckenooghe A. Symptomatic Dengue Disease in Five Southeast Asian Countries: Epidemiological Evidence from a Dengue Vaccine Trial. PLoS Negl Trop Dis. 2016 Aug 17;10(8):e0004918. doi: 10.1371/journal.pntd.0004918. eCollection 2016 Aug. PMID 27532617
- [Result] Olivera-Botello G, Coudeville L, Fanouillere K, Guy B, Chambonneau L, Noriega F, Jackson N; CYD-TDV Vaccine Trial Group. Tetravalent Dengue Vaccine Reduces Symptomatic and Asymptomatic Dengue Virus Infections in Healthy Children and Adolescents Aged 2-16 Years in Asia and Latin America. J Infect Dis. 2016 Oct 1;214(7):994-1000. doi: 10.1093/infdis/jiw297. Epub 2016 Jul 14. PMID 27418050
- [Result] Coudeville L, Baurin N, L'Azou M, Guy B. Potential impact of dengue vaccination: Insights from two large-scale phase III trials with a tetravalent dengue vaccine. Vaccine. 2016 Dec 7;34(50):6426-6435. doi: 10.1016/j.vaccine.2016.08.050. Epub 2016 Sep 3. PMID 27601343
- [Result] Sridhar S, Luedtke A, Langevin E, Zhu M, Bonaparte M, Machabert T, Savarino S, Zambrano B, Moureau A, Khromava A, Moodie Z, Westling T, Mascarenas C, Frago C, Cortes M, Chansinghakul D, Noriega F, Bouckenooghe A, Chen J, Ng SP, Gilbert PB, Gurunathan S, DiazGranados CA. Effect of Dengue Serostatus on Dengue Vaccine Safety and Efficacy. N Engl J Med. 2018 Jul 26;379(4):327-340. doi: 10.1056/NEJMoa1800820. Epub 2018 Jun 13. PMID 29897841
- [Derived] Savarino SJ, Bonaparte M, Wang H, Dayan GH, Forrat R, Zhu M, Hodge S, Ataman-Onal Y, DiazGranados CA. Accuracy and efficacy of pre-dengue vaccination screening for previous dengue infection with a new dengue rapid diagnostic test: a retrospective analysis of phase 3 efficacy trials. Lancet Microbe. 2022 Jun;3(6):e427-e434. doi: 10.1016/S2666-5247(22)00033-7. Epub 2022 May 4. PMID 35659904
- [Derived] Laydon DJ, Dorigatti I, Hinsley WR, Nedjati-Gilani G, Coudeville L, Ferguson NM. Efficacy profile of the CYD-TDV dengue vaccine revealed by Bayesian survival analysis of individual-level phase III data. Elife. 2021 Jul 2;10:e65131. doi: 10.7554/eLife.65131. PMID 34219653
- [Derived] Henein S, Adams C, Bonaparte M, Moser JM, Munteanu A, Baric R, de Silva AM. Dengue vaccine breakthrough infections reveal properties of neutralizing antibodies linked to protection. J Clin Invest. 2021 Jul 1;131(13):e147066. doi: 10.1172/JCI147066. PMID 34003796
- [Derived] Forrat R, Dayan GH, DiazGranados CA, Bonaparte M, Laot T, Capeding MR, Sanchez L, Coronel DL, Reynales H, Chansinghakul D, Hadinegoro SRS, Perroud AP, Frago C, Zambrano B, Machabert T, Wu Y, Luedtke A, Price B, Vigne C, Haney O, Savarino SJ, Bouckenooghe A, Noriega F. Analysis of Hospitalized and Severe Dengue Cases Over the 6 years of Follow-up of the Tetravalent Dengue Vaccine (CYD-TDV) Efficacy Trials in Asia and Latin America. Clin Infect Dis. 2021 Sep 15;73(6):1003-1012. doi: 10.1093/cid/ciab288. PMID 33822015
- [Derived] DiazGranados CA, Bonaparte M, Wang H, Zhu M, Lustig Y, Schwartz E, Forrat R, Dayan GH, Hodge S, Ataman-Onal Y, Savarino SJ. Accuracy and efficacy of pre-dengue vaccination screening for previous dengue infection with five commercially available immunoassays: a retrospective analysis of phase 3 efficacy trials. Lancet Infect Dis. 2021 Apr;21(4):529-536. doi: 10.1016/S1473-3099(20)30695-2. Epub 2020 Nov 16. PMID 33212068
- [Derived] Plennevaux E, Moureau A, Arredondo-Garcia JL, Villar L, Pitisuttithum P, Tran NH, Bonaparte M, Chansinghakul D, Coronel DL, L'Azou M, Ochiai RL, Toh ML, Noriega F, Bouckenooghe A. Impact of Dengue Vaccination on Serological Diagnosis: Insights From Phase III Dengue Vaccine Efficacy Trials. Clin Infect Dis. 2018 Apr 3;66(8):1164-1172. doi: 10.1093/cid/cix966. PMID 29300876
- [Derived] Rabaa MA, Girerd-Chambaz Y, Duong Thi Hue K, Vu Tuan T, Wills B, Bonaparte M, van der Vliet D, Langevin E, Cortes M, Zambrano B, Dunod C, Wartel-Tram A, Jackson N, Simmons CP. Genetic epidemiology of dengue viruses in phase III trials of the CYD tetravalent dengue vaccine and implications for efficacy. Elife. 2017 Sep 5;6:e24196. doi: 10.7554/eLife.24196. PMID 28871961
- [Derived] Harenberg A, de Montfort A, Jantet-Blaudez F, Bonaparte M, Boudet F, Saville M, Jackson N, Guy B. Cytokine Profile of Children Hospitalized with Virologically-Confirmed Dengue during Two Phase III Vaccine Efficacy Trials. PLoS Negl Trop Dis. 2016 Jul 26;10(7):e0004830. doi: 10.1371/journal.pntd.0004830. eCollection 2016 Jul. PMID 27459266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 03 June 2011 to 01 December 2011 at 9 sites in Indonesia, 5 in Malaysia, 3 in Thailand, 5 in Philippines, and 2 in Vietnam.
Pre-assignment Details: A total of 10275 participants were enrolled; all but one met all of the inclusion criteria and none of the exclusion criteria. Three participants were not vaccinated and were excluded from the Full Analysis Set for Efficacy and the Safety Analysis Set.
Groups:
- CYD Dengue Vaccine Group: Participants received 3 doses of CYD dengue vaccine; one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (or a total duration of up to 72 months).
- Placebo Group: Participants received 3 doses of placebo matched to vaccine; one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (or a total duration of up to 72 months).
Period: Vaccination Phase (Up to 25 Months)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 6851 | 3424
Completed | 6797 | 3397
Not Completed | 54 | 27
Not completed — Withdrawal by Subject | 40 | 23
Not completed — Protocol Violation | 5 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Serious adverse event | 4 | 1
Period: Surveillance Expansion Period
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 6797 | 3397
Completed | 6595 | 3279
Not Completed | 202 | 118
Not completed — Withdrawal by Subject | 180 | 105
Not completed — Protocol Violation | 9 | 1
Not completed — Lost to Follow-up | 10 | 8
Not completed — Serious adverse event | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Participants received 3 doses of placebo vaccine, one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (or a total duration of up to 72 months).
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 6851 | 3424 | 10275
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6851 | 3424 | 10275
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 8.8 (3.45) | 8.8 (3.42) | 8.8 (3.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3524 | 1767 | 5291
  Male | 3327 | 1657 | 4984
Region of Enrollment [Count of Participants; unit: Participants]
  Philippines | 2335 | 1166 | 3501
  Malaysia | 937 | 464 | 1401
  Indonesia | 1246 | 624 | 1870
  Thailand | 778 | 392 | 1170
  Vietnam | 1555 | 778 | 2333

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptomatic Virologically Confirmed Dengue (VCD) Cases Due to Any Serotype During the Active Phase Post-dose 3 Following Injection (Inj.) With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as occurrence of acute febrile illness (temperature >=38°C on at least 2 consecutive days) and confirmation of dengue virus infection by dengue reverse transcriptase polymerase chain reaction and/or dengue NS protein 1 antigen enzyme-linked immunosorbent assay. Vaccine efficacy was defined as 1 minus the ratio of density incidence due to any serotype after at least 1 dose in the CYD Dengue Vaccine Group over the density incidence of the Placebo Vaccine Group.
Time Frame: 28 days and up to 13 months post-dose 3
Population: Number of symptomatic VCD cases were assessed in the Per-Protocol Analysis Set for Efficacy
Measure: Number; unit: Cases
Groups:
- CYD Dengue Vaccine Group: Participants were to receive 3 doses of CYD dengue vaccine; one each at 0, 6, and 12 months.
- Placebo Group: Participants were to receive 3 doses of placebo vaccine, one each at 0, 6, and 12 months.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6709 | 3350
Cases | 117 | 133
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; The statistical methodology was based on the use of the two-sided 95% confidence interval (CI) of the vaccine efficacy (expressed in %). The CI was calculated using the exact method conditional on the total number of cases in both groups (exact method by Breslow & Day). The vaccine efficacy of the CYD dengue vaccine was considered significant if the lower bound of its 95% CI was greater than 25%; Test type: Superiority or Other; Vaccine efficacy = 56.5, 95% CI 2-sided [43.8 to 66.4]

2. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each Serotype With the Parental Dengue Virus Strain Before and Following Injection With Either CYD Dengue Tetravalent Vaccine or a Placebo
Description: Geometric mean titers against each of the 4 serotypes of dengue virus strains were assessed using the plaque reduction neutralization test (PRNT) in a pre-defined subset of participants.
Time Frame: Pre-injection 1, 28 days post Injections 2 and 3, 13 months (Visit 07) and 60 months (Visit 12) post-injection 3
Population: Antibody titers against each dengue virus serotype strain were assessed in Full Analysis Set for Immunogenicity(FASI),which included a subset of participants who received at least one dose of vaccine and had a blood sample drawn and result available after the dose. Here,'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Groups:
- CYD Dengue Vaccine Group: Subset of participants who received at least one dose of CYD Dengue vaccine.
- Placebo Group: Subset of participants who received at least one dose of the placebo vaccine.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 1323 | 660
Titers (1/dilution)
  Dengue virus Serotype 1; Pre-Inj. 1: number analyzed (Participants) | 1309 | 655
  Dengue virus Serotype 1; Pre-Inj. 1 | 38.3 [33.8 to 43.5] | 42.1 [35 to 50.6]
  Dengue virus Serotype 1; Post Inj. 2: number analyzed (Participants) | 1317 | 654
  Dengue virus Serotype 1; Post Inj. 2 | 153 [137 to 170] | 46.1 [38.2 to 55.7]
  Dengue virus Serotype 1; Post Inj. 3: number analyzed (Participants) | 1316 | 657
  Dengue virus Serotype 1; Post Inj. 3 | 166 [150 to 183] | 46.6 [38.7 to 56.1]
  Dengue virus Serotype 1; Year 1 Post Inj. 3 (V 07): number analyzed (Participants) | 1290 | 634
  Dengue virus Serotype 1; Year 1 Post Inj. 3 (V 07) | 105 [92.8 to 119] | 57.2 [46.9 to 69.8]
  Dengue virus Serotype 1; Year 5 Post Inj. 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 1; Year 5 Post Inj. 3 (V 12) | 81.2 [72.5 to 91.0] | 77.6 [65.4 to 92.2]
  Dengue virus Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 1313 | 654
  Dengue virus Serotype 2; Pre-Inj. 1 | 55.3 [48.7 to 62.9] | 62.1 [51.7 to 74.7]
  Dengue virus Serotype 2; Post Inj. 2: number analyzed (Participants) | 1316 | 655
  Dengue virus Serotype 2; Post Inj. 2 | 360 [329 to 394] | 69.5 [57.7 to 83.6]
  Dengue virus Serotype 2; Post Inj. 3: number analyzed (Participants) | 1314 | 657
  Dengue virus Serotype 2; Post Inj. 3 | 355 [327 to 386] | 68.5 [57.1 to 82.2]
  Dengue virus Serotype 2; Year 1 Post-Inj. 3 (V 07): number analyzed (Participants) | 1298 | 640
  Dengue virus Serotype 2; Year 1 Post-Inj. 3 (V 07) | 194 [175 to 214] | 78.1 [64.8 to 94.0]
  Dengue virus Serotype 2; Year 5 Post-Inj. 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 2; Year 5 Post-Inj. 3 (V 12) | 144 [130 to 160] | 102 [86.8 to 120]
  Dengue virus Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 1307 | 650
  Dengue virus Serotype 3; Pre-Inj. 1 | 40.1 [35.6 to 45.1] | 40.7 [34.5 to 48]
  Dengue virus Serotype 3; Post Inj. 2: number analyzed (Participants) | 1313 | 656
  Dengue virus Serotype 3; Post Inj. 2 | 203 [184 to 223] | 40.8 [34.6 to 48.1]
  Dengue virus Serotype 3; Post Inj. 3: number analyzed (Participants) | 1314 | 657
  Dengue virus Serotype 3; Post Inj. 3 | 207 [189 to 226] | 42.5 [36.2 to 49.9]
  Dengue virus Serotype 3; Year 1 Post Inj. 3 (V 07): number analyzed (Participants) | 1298 | 639
  Dengue virus Serotype 3; Year 1 Post Inj. 3 (V 07) | 186 [168 to 206] | 62.1 [51.8 to 74.6]
  Dengue virus Serotype 3; Year 5 Post Inj. 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 3; Year 5 Post Inj. 3 (V 12) | 120 [108 to 133] | 76.2 [65.3 to 89.0]
  Dengue virus Serotype 4; Pre Inj. 1: number analyzed (Participants) | 1313 | 653
  Dengue virus Serotype 4; Pre Inj. 1 | 25.3 [22.9 to 28] | 26.2 [22.6 to 30.3]
  Dengue virus Serotype 4; Post Inj. 2: number analyzed (Participants) | 1318 | 655
  Dengue virus Serotype 4; Post Inj. 2 | 151 [139 to 163] | 24.4 [21.3 to 28.1]
  Dengue virus Serotype 4; Post Inj. 3: number analyzed (Participants) | 1315 | 657
  Dengue virus Serotype 4; Post Inj. 3 | 151 [141 to 162] | 26.0 [22.6 to 29.8]
  Dengue virus Serotype 4; Year 1 Post Inj. 3 (V 07): number analyzed (Participants) | 1293 | 621
  Dengue virus Serotype 4; Year 1 Post Inj. 3 (V 07) | 85.5 [78.5 to 93] | 26.0 [22.4 to 30.3]
  Dengue virus Serotype 4; Year 5 Post Inj. 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 4; Year 5 Post Inj. 3 (V 12) | 65.7 [60.3 to 71.6] | 40.1 [34.8 to 46.1]

3. Secondary Outcome: Percentage of Participants With Antibody Titers >= 10 1/Dilution (1/Dil) Against Each Dengue Virus Serotype Strain Before and Following Inj. With CYD Dengue Vaccine or Placebo
Description: Percentage of participants with antibody titers >= 10 (1/Dil) against each serotypes of the dengue virus strains were assessed using PRNT in a pre-defined subset of participants.
Time Frame: Pre-injection 1, 28 days post Injections 2 and 3, 13 months (V 07) and 60 months (V 12) post-injection 3
Population: Antibody titers against each dengue virus serotype strain were assessed in FASI, which included a subset of participants who received at least one dose of vaccine and had a blood sample drawn and result available after the dose. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo Group: Subset of participants who received at least one dose of placebo vaccine
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 1323 | 660
Percentage of participants
  Dengue virus Serotype 1; Pre-Inj. 1: number analyzed (Participants) | 1309 | 655
  Dengue virus Serotype 1; Pre-Inj. 1 | 52.0 | 51.3
  Dengue virus Serotype 1; Post Inj. 2: number analyzed (Participants) | 1317 | 654
  Dengue virus Serotype 1; Post Inj. 2 | 88.9 | 54.4
  Dengue virus Serotype 1; Post-Inj. 3: number analyzed (Participants) | 1316 | 657
  Dengue virus Serotype 1; Post-Inj. 3 | 94.0 | 55.4
  Dengue virus Serotype 1; Year 1 Post-Inj. 3 (V 07): number analyzed (Participants) | 1290 | 634
  Dengue virus Serotype 1; Year 1 Post-Inj. 3 (V 07) | 79.8 | 55.7
  Dengue virus Serotype 1; Year 5 Post-Inj 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 1; Year 5 Post-Inj 3 (V 12) | 76.2 | 70.0
  Dengue virus Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 1313 | 654
  Dengue virus Serotype 2; Pre-Inj. 1 | 58.0 | 59.3
  Dengue virus Serotype 2; Post-Inj. 2: number analyzed (Participants) | 1316 | 655
  Dengue virus Serotype 2; Post-Inj. 2 | 97.3 | 62.4
  Dengue virus Serotype 2; Post-Inj. 3: number analyzed (Participants) | 1314 | 657
  Dengue virus Serotype 2; Post-Inj. 3 | 98.7 | 61.8
  Dengue virus Serotype 2; Year 1 Post-Inj. 3 (V 07): number analyzed (Participants) | 1298 | 640
  Dengue virus Serotype 2; Year 1 Post-Inj. 3 (V 07) | 92.0 | 65.8
  Dengue virus Serotype 2; Year 5 Post-inj 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 2; Year 5 Post-inj 3 (V 12) | 86 | 75.2
  Dengue virus Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 1307 | 650
  Dengue virus Serotype 3; Pre-Inj. 1 | 56.8 | 59.4
  Dengue virus Serotype 3; Post-Inj. 2: number analyzed (Participants) | 1313 | 656
  Dengue virus Serotype 3; Post-Inj. 2 | 95.7 | 60.2
  Dengue virus Serotype 3; Post-Inj. 3: number analyzed (Participants) | 1314 | 657
  Dengue virus Serotype 3; Post-Inj. 3 | 97.0 | 61.0
  Dengue virus Serotype 3; Year 1 Post-Inj. 3 (V 07): number analyzed (Participants) | 1298 | 639
  Dengue virus Serotype 3; Year 1 Post-Inj. 3 (V 07) | 93.6 | 62.6
  Dengue virus Serotype 3; Year5 Post-Inj. 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 3; Year5 Post-Inj. 3 (V 12) | 87.4 | 75.6
  Dengue virus Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 1313 | 653
  Dengue virus Serotype 4; Pre-Inj. 1 | 51.6 | 50.7
  Dengue virus Serotype 4; Post-Inj. 2: number analyzed (Participants) | 1318 | 655
  Dengue virus Serotype 4; Post-Inj. 2 | 95.1 | 51.8
  Dengue virus Serotype 4; Post-Inj. 3: number analyzed (Participants) | 1315 | 657
  Dengue virus Serotype 4; Post-Inj. 3 | 97.0 | 53.9
  Dengue virus Serotype 4; Year 1 Post-Inj 3 (V 07): number analyzed (Participants) | 1293 | 621
  Dengue virus Serotype 4; Year 1 Post-Inj 3 (V 07) | 89.4 | 50.6
  Dengue virus Serotype 4; Year 5 Post-Inj 3 (V 12): number analyzed (Participants) | 1275 | 640
  Dengue virus Serotype 4; Year 5 Post-Inj 3 (V 12) | 83.8 | 65.0

4. Secondary Outcome: Number of Symptomatic VCD Cases Due to Any Serotype Occurring 28 Days Post-dose 1 Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as occurrence of acute febrile illness (temperature >= 38°C on at least 2 consecutive days) and confirmation of dengue virus infection by dengue reverse transcriptase polymerase chain reaction and/or dengue NS1 enzyme-linked immunosorbent assay. Vaccine efficacy was defined as 1 minus the ratio of density incidence due to any serotype after at least 1 dose in the CYD Dengue Vaccine Group over the density incidence of the Placebo Vaccine Group.
Time Frame: 28 days post-injection 1 and up to 13 months post-injection 3
Population: Number of symptomatic VCD cases were assessed in the Full Analysis Set for Efficacy, which included participants who received at least 1 dose of study vaccine.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6848 | 3424
Cases | 276 | 302
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; The statistical methodology was based on the use of the two-sided 95% CI of the vaccine efficacy (expressed in %) calculated using the exact method conditional on the total number of cases in both groups; Test type: Superiority or Other; Vaccine Efficacy = 55.4, 95% CI 2-sided [47.3 to 62.3]

5. Secondary Outcome: Number of Symptomatic VCD Cases Due to Any Serotype 28 Days Post-dose 2 Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: as for outcome 4
Time Frame: 28 days post-injection 2 and up to 13 months post-injection 3
Population: Number of symptomatic VCD cases were assessed in the Other Efficacy Analysis Set, which included participants who received at least 2 doses of study vaccine.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6793 | 3397
Cases | 205 | 238
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Vaccine Efficacy = 57.9, 95% CI 2-sided [49.0 to 65.2]

6. Secondary Outcome: Number of Symptomatic VCD Cases Due to Any Serotype During the Active Phase in Either CYD Dengue Vaccine or Placebo Group
Description: Symptomatic VCD cases were defined as occurrence of acute febrile illness (temperature >=38°C on at least 2 consecutive days) and confirmation of dengue virus infection by dengue reverse transcriptase polymerase chain reaction and/or dengue NS1 enzyme-linked immunosorbent assay. Vaccine efficacy was defined as 1 minus the ratio of density incidence due to any serotype after at least 1 dose in the CYD Dengue Vaccine Group over the density incidence of the Placebo Vaccine Group.
Time Frame: Day 0 up to 13 months post-injection 3
Population: Number of symptomatic VCD cases were assessed in the Full Analysis Set for Efficacy, which included all participants who received at least 1 injection.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6848 | 3424
Cases | 286 | 309
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Vaccine Efficacy = 54.8, 95% CI 2-sided [46.8 to 61.7]

7. Secondary Outcome: Number of Symptomatic VCD Cases Meeting 1997 WHO Criteria Throughout the Trial Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Dengue hemorrhagic fever cases were defined as number of participants with at least one symptomatic VCD episode meeting the 1997 WHO criteria.
  (a) Fever: acute onset, high (>= 38°C) and continuous, lasting 2 to 7 days and (b) any of the pre-listed hemorrhagic manifestations and laboratory findings of thrombocytopenia (platelet <=100 x 109/L) and plasma leakage as shown by hemoconcentation (hematocrit increased by 20% or more) or pleural effusion (seen on CXR) and/or ascites and/or hypoaluminemia. The first two clinical criteria plus thrombocytopenia and signs of plasma leakage are enough to establish a clinical diagnosis of DHF. Dengue hemorrhagic fever was graded as follows: Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test; Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participants, usually in the form of skin and/or other hemorrhage.
Time Frame: Day 0 to the end of study (up to 72 months)
Population: Number of WHO dengue hemorrhagic fever cases were assessed in the Safety Analysis Set, which included all participants who received at least one dose of study vaccine. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6848 | 3424
Cases
  Due to Any of the 4 Serotypes: Any Grade: number analyzed (Participants) | 6745 | 3369
  Due to Any of the 4 Serotypes: Any Grade | 55 | 41
  Due to Any of the 4 Serotypes: Grade I: number analyzed (Participants) | 6745 | 3369
  Due to Any of the 4 Serotypes: Grade I | 14 | 9
  Due to Any of the 4 Serotypes: Grade II: number analyzed (Participants) | 6745 | 3369
  Due to Any of the 4 Serotypes: Grade II | 37 | 29
  Due to Any of the 4 Serotypes: Grade III: number analyzed (Participants) | 6745 | 3369
  Due to Any of the 4 Serotypes: Grade III | 4 | 3
  Due to Any of the 4 Serotypes: Grade IV: number analyzed (Participants) | 6745 | 3369
  Due to Any of the 4 Serotypes: Grade IV | 0 | 0

8. Secondary Outcome: Number of Symptomatic VCD Cases Meeting 1997 WHO Criteria During the Surveillance Expansion Period Due to Any Serotype Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: The 1997 WHO criteria are: a) Fever: acute onset, high (>= 38°C) and continuous, for 2 to 7 days and (b) any of the following: thrombocytopenia (platelet <=100 x 109/L) and plasma leakage as shown by hematocrit increased by 20% or more or pleural effusion and/or ascites and/or hypoaluminemia. The first two clinical criteria plus thrombocytopenia and signs of plasma leakage are enough to establish diagnosis of DHF. Dengue hemorrhagic fever was graded as follows:Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test; Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participant,usually in the form of skin and/or other hemorrhages; Grade III: Circulatory failure manifested by rapid and weak pulse, narrowing of pulse pressure (20 mmHg or less) or hypotension, with the presence of cold clammy skin and restlessness; and Grade IV: Profound shock with undetectable blood pressure and pulse.
Time Frame: From consent to participate int the Surveillance Expansion Period to 60 months post-injection 3 (up to Month 72)
Population: Number of WHO dengue hemorrhagic fever cases were assessed in the Full Analysis Set for Surveillance Expansion Period, which included all participants who received at least 1 injection and accepted to be included in the Surveillance Expansion Period.
Measure: Number; unit: Cases
Groups:
- Placebo Group: Participant were to receive 3 doses of placebo vaccine, one each at 0, 6, and 12 months.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6327 | 3138
Cases
  Due to Any of the 4 Serotypes: Any Grade | 19 | 12
  Due to Any of the 4 Serotypes: Grade I | 5 | 3
  Due to Any of the 4 Serotypes: Grade II | 11 | 8
  Due to Any of the 4 Serotypes: Grade III | 3 | 1
  Due to Any of the 4 Serotypes: Grade IV | 0 | 0

9. Secondary Outcome: Number of Clinically Severe VCD Cases Throughout the Trial Due to Any Serotype Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: The severity of VCD cases was assessed by an IDMC based on a medical review of cases and any of the following criteria:1) Platelet count <=100000 μl and bleeding (tourniquet, petechiae or any bleeding) plus plasma leakage 2) Shock (pulse pressure <= 20 mmHg in a child, or hypotension [<= 90 mmHg] with tachycardia, weak pulse and poor perfusion) 3) Bleeding requiring blood transfusion 4) Encephalopathy i.e. Unconsciousness or poor conscious state or fitting not attributable to simple febrile convulsion or focal neurological signs. Poor conscious state or unconsciousness must be supported by GCS score 5) Liver impairment (AST >1000 IU/L or PT INR >1.5) excluding other causes of viral hepatitis 6) Impaired kidney function (serum creatinine >= 1.5 mg/dL) 7) Myocarditis, pericarditis or clinical heart failure supported by CXR, echocardiography, ECG or cardiac enzymes.
Time Frame: Day 0 to the end of study (up to 72 months)
Population: Number of clinically severe VCD cases were assessed in the Safety Analysis Set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6745 | 3369
Cases | 61 | 41

10. Secondary Outcome: Number of Clinically Severe VCD Cases During the Surveillance Expansion Period Due to Any Serotype Following Inj. With Either CYD Dengue Vaccine or a Placebo
Description: The severity of VCD cases was assessed by an IDMC based on a medical review of cases and any of the following criteria:1) Platelet count <=100000μl and bleeding (tourniquet, petechiae or any bleeding) plus plasma leakage 2) Shock (pulse pressure <= 20mmHg in a child, or hypotension [<= 90 mmHg] with tachycardia, weak pulse and poor perfusion) 3) Bleeding requiring blood transfusion 4) Encephalopathy i.e. Unconsciousness or poor conscious state or fitting not attributable to simple febrile convulsion or focal neurological signs. Poor conscious state or unconsciousness must be supported by GCS score 5) Liver impairment (AST >1000 IU/L or PT INR >1.5) excluding other causes of viral hepatitis 6) Impaired kidney function (serum creatinine >= 1.5 mg/dL) 7) Myocarditis, pericarditis or clinical heart failure supported by CXR, echocardiography, ECG or cardiac enzymes.
Time Frame: From consent to participate in the Surveillance Expansion Period to 60 months post-injection 3 (up to Month 72)
Population: Number of clinically severe VCD cases were assessed in the Full Analysis Set for SEP.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6327 | 3138
Cases | 21 | 12

11. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions Following Any and Each Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Grade 3 reactions (2-11 years): Pain, Incapacitating, unable to perform usual activities; Erythema and Swelling, >= 50 mm. Grade 3 Solicited injection site reactions (12-14 years): Pain, Significant, prevents daily activity; Erythema and Swelling, >100 mm.
Time Frame: Within 7 days after injection
Population: Solicited injection site reactions were assessed in a subset of the Safety Analysis Set, which included all participants who received at least one dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 1334 | 663
participants
  Injection-site Pain (Post any injection): number analyzed (Participants) | 1332 | 663
  Injection-site Pain (Post any injection) | 614 | 275
  Injection-site Erythema (Post-any injection): number analyzed (Participants) | 1332 | 663
  Injection-site Erythema (Post-any injection) | 107 | 52
  Injection-site Swelling (Post any injection): number analyzed (Participants) | 1332 | 663
  Injection-site Swelling (Post any injection) | 68 | 33
  Injection-site Pain (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Injection-site Pain (Post-injection 1) | 406 | 196
  Grade 3 Injection-site Pain (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Grade 3 Injection-site Pain (Post-injection 1) | 1 | 0
  Injection-site Erythema (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Injection-site Erythema (Post-injection 1) | 63 | 35
  Grade 3 Injection-site Erythema (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Grade 3 Injection-site Erythema (Post-injection 1) | 0 | 0
  Injection-site Swelling (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Injection-site Swelling (Post-injection 1) | 40 | 19
  Grade 3 Injection-site Swelling (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Grade 3 Injection-site Swelling (Post-injection 1) | 0 | 0
  Injection-site Pain (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Injection-site Pain (Post-injection 2) | 303 | 135
  Grade 3 Injection-site Pain (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Grade 3 Injection-site Pain (Post-injection 2) | 0 | 0
  Injection-site Erythema (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Injection-site Erythema (Post-injection 2) | 43 | 20
  Grade 3 Injection-site Erythema (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Grade 3 Injection-site Erythema (Post-injection 2) | 0 | 0
  Injection-site Swelling (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Injection-site Swelling (Post-injection 2) | 25 | 7
  Grade 3 Injection-site Swelling (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Grade 3 Injection-site Swelling (Post-injection 2) | 0 | 0
  Injection-site Pain (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Injection-site Pain (Post-injection 3) | 283 | 118
  Grade 3 Injection-site Pain (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Grade 3 Injection-site Pain (Post-injection 3) | 0 | 0
  Injection-site Erythema (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Injection-site Erythema (Post-injection 3) | 36 | 16
  Grade 3 Injection-site Erythema (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Grade 3 Injection-site Erythema (Post-injection 3) | 0 | 1
  Injection-site Swelling (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Injection-site Swelling (Post-injection 3) | 19 | 10
  Grade 3 Injection-site Swelling (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Grade 3 Injection-site Swelling (Post-injection 3) | 0 | 0

12. Secondary Outcome: Number of Participants With Systemic Reactions Following Any and Each Inj. With Either CYD Dengue Vaccine or a Placebo
Description: Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Asthenia. Grade 3 reactions: Fever, >= 39°C; Headache, Malaise, Myalgia, and Asthenia, Significant, prevents daily activity.
Time Frame: Within 14 days after injection
Population: Solicited systemic reactions were assessed in a subset of the Safety Analysis Set, which included all participants who received at least one dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 1334 | 663
participants
  Fever (Post any injection): number analyzed (Participants) | 1332 | 663
  Fever (Post any injection) | 248 | 118
  Headache (Post any injection): number analyzed (Participants) | 1332 | 663
  Headache (Post any injection) | 562 | 259
  Malaise (Post any injection): number analyzed (Participants) | 1332 | 663
  Malaise (Post any injection) | 476 | 239
  Myalgia (Post any injection): number analyzed (Participants) | 1332 | 663
  Myalgia (Post any injection) | 414 | 197
  Asthenia (Post any injection): number analyzed (Participants) | 1332 | 663
  Asthenia (Post any injection) | 378 | 167
  Fever (Post-injection 1): number analyzed (Participants) | 1330 | 663
  Fever (Post-injection 1) | 103 | 45
  Grade 3 Fever (Post-injection 1): number analyzed (Participants) | 1330 | 663
  Grade 3 Fever (Post-injection 1) | 18 | 7
  Headache (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Headache (Post-injection 1) | 387 | 168
  Grade 3 Headache (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Grade 3 Headache (Post-injection 1) | 7 | 6
  Malaise (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Malaise (Post-injection 1) | 312 | 148
  Grade 3 Malaise (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Grade 3 Malaise (Post-injection 1) | 7 | 4
  Myalgia (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Myalgia (Post-injection 1) | 255 | 124
  Grade 3 Myalgia (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Grade 3 Myalgia (Post-injection 1) | 2 | 2
  Asthenia (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Asthenia (Post-injection 1) | 229 | 97
  Grade 3 Asthenia (Post-injection 1): number analyzed (Participants) | 1332 | 663
  Grade 3 Asthenia (Post-injection 1) | 5 | 5
  Fever (Post-injection 2): number analyzed (Participants) | 1320 | 657
  Fever (Post-injection 2) | 90 | 44
  Grade 3 Fever (Post-injection 2): number analyzed (Participants) | 1320 | 657
  Grade 3 Fever (Post-injection 2) | 19 | 9
  Headache (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Headache (Post-injection 2) | 247 | 118
  Grade 3 Headache (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Grade 3 Headache (Post-injection 2) | 12 | 3
  Malaise (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Malaise (Post-injection 2) | 192 | 100
  Grade 3 Malaise (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Grade 3 Malaise (Post-injection 2) | 6 | 4
  Myalgia (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Myalgia (Post-injection 2) | 174 | 92
  Grade 3 Myalgia (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Grade 3 Myalgia (Post-injection 2) | 3 | 0
  Asthenia (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Asthenia (Post-injection 2) | 158 | 74
  Grade 3 Asthenia (Post-injection 2): number analyzed (Participants) | 1319 | 658
  Grade 3 Asthenia (Post-injection 2) | 5 | 6
  Fever (Post-injection 3): number analyzed (Participants) | 1309 | 654
  Fever (Post-injection 3) | 76 | 39
  Grade 3 Fever (Post-injection 3): number analyzed (Participants) | 1309 | 654
  Grade 3 Fever (Post-injection 3) | 16 | 2
  Headache (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Headache (Post-injection 3) | 219 | 113
  Grade 3 Headache (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Grade 3 Headache (Post-injection 3) | 6 | 1
  Malaise (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Malaise (Post-injection 3) | 183 | 104
  Grade 3 Malaise (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Grade 3 Malaise (Post-injection 3) | 7 | 1
  Myalgia (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Myalgia (Post-injection 3) | 156 | 76
  Grade 3 Myalgia (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Grade 3 Myalgia (Post-injection 3) | 3 | 0
  Asthenia (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Asthenia (Post-injection 3) | 142 | 73
  Grade 3 Asthenia (Post-injection 3): number analyzed (Participants) | 1313 | 654
  Grade 3 Asthenia (Post-injection 3) | 4 | 2

13. Secondary Outcome: Number of Hospitalized VCD Cases Throughout the Trial Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Hospitalized VCD cases were defined as VCD confirmed by dengue RT-PCR and/or dengue NS1 ELISA in participants with acute febrile illness (temperature >=38°C on at least 2 consecutive days) requiring hospitalization.
Time Frame: Day 0 to the end of study (up to 72 months)
Population: Number of hospitalized dengue hemorrhagic fever cases were assessed in the Safety Analysis Set. Here, 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Cases
Groups:
- CYD Dengue Vaccine Group: Participants were to receive 3 doses of CYD dengue vaccine; one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (up to 72 months).
- Placebo Group: Participants were to receive 3 doses of placebo matched to vaccine; one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (up to 72 months).
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6745 | 3369
Cases | 210 | 154

14. Secondary Outcome: Number of Hospitalized VCD Cases During the Surveillance Expansion Period Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Hospitalized VCD cases were defined as VCD confirmed by dengue RT-PCR and/or dengue NS1 ELISA in participants with acute febrile illness (temperature >= 38°C on at least 2 consecutive days) requiring hospitalization.
Time Frame: From consent to participate in the Surveillance Expansion Period to 60 months post-injection 3 (up to Month 72)
Population: Number of hospitalized dengue hemorrhagic fever cases were assessed in the Safety Analysis Set.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 6848 | 3424
Cases | 74 | 48

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to 60 months post-injection 3 (up to 72 months).
Description: All the vaccinated participants were assessed for SAE during the trial. Non-serious adverse events included solicited injection-site (within 7 days after injection) and solicited systemic reactions (within 14 days after injection), as well as unsolicited non-serious adverse events (within 28 days after injection). These events were assessed in a subset of participants from each group, who had received at least 1 dose of study vaccine.
Groups:
- Placebo Group: Participants were to receive 3 doses of placebo vaccine; one each at 0, 6, and 12 months.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 10/6848 | 4/3424
Serious Adverse Events (participants affected / at risk) | 947/6848 | 552/3424
Other Adverse Events (participants affected / at risk) | 942/1334 | 453/663
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=6848) | Placebo Group (N=3424)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia Of Pregnancy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Rheumatic Heart Disease (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (2) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Duchenne Muscular Dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Familial Periodic Paralysis (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Fibrous Dysplasia Of Bone (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Odontogenic Cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular Disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 3 (3) | 0 (0)
Choroidal Dystrophy (Eye disorders) | 1 (1) | 0 (0)
Corneal Oedema (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Caecitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 2 (2)
Enteritis (Gastrointestinal disorders) | 5 (5) | 1 (2)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 9 (9) | 3 (3)
Gastritis (Gastrointestinal disorders) | 31 (32) | 14 (16)
Gastrointestinal Disorder (Gastrointestinal disorders) | 9 (10) | 5 (5)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary Gland Calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary Gland Mucocoele (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tooth Development Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth Impacted (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 1 (1) | 0 (0)
Hernia Obstructive (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy To Arthropod Bite (Immune system disorders) | 1 (1) | 1 (1)
Allergy To Arthropod Sting (Immune system disorders) | 4 (4) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 3 (3) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 1 (1) | 2 (2)
Drug Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Food Allergy (Immune system disorders) | 5 (5) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2)
Abscess Limb (Infections and infestations) | 4 (4) | 0 (0)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0)
Abscess Of External Auditory Meatus (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Acute Tonsillitis (Infections and infestations) | 7 (7) | 2 (2)
Adenoiditis (Infections and infestations) | 4 (4) | 1 (1)
Amoebiasis (Infections and infestations) | 9 (9) | 4 (4)
Amoebic Dysentery (Infections and infestations) | 3 (3) | 2 (2)
Anal Abscess (Infections and infestations) | 0 (0) | 2 (2)
Appendiceal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 33 (33) | 27 (27)
Appendicitis Perforated (Infections and infestations) | 5 (5) | 4 (4)
Bacterial Diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Infection (Infections and infestations) | 2 (2) | 1 (1)
Bartholin's Abscess (Infections and infestations) | 2 (3) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 16 (16) | 6 (8)
Bronchitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 8 (8) | 1 (1)
Brucellosis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 7 (7) | 3 (3)
Chikungunya Virus Infection (Infections and infestations) | 2 (2) | 0 (0)
Chronic Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 3 (3) | 0 (0)
Dengue Fever (Infections and infestations) | 238 (241) | 158 (167)
Diarrhoea Infectious (Infections and infestations) | 3 (3) | 5 (5)
Disseminated Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis Viral (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 3 (3) | 0 (0)
Gastritis Bacterial (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 53 (64) | 40 (43)
Gastroenteritis Bacterial (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 3 (3) | 1 (1)
Gastrointestinal Bacterial Infection (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 6 (6) | 5 (5)
Groin Abscess (Infections and infestations) | 2 (2) | 0 (0)
Hiv Infection (Infections and infestations) | 1 (1) | 0 (0)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis A (Infections and infestations) | 2 (2) | 1 (1)
Hepatitis Viral (Infections and infestations) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Infection In An Immunocompromised Host (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 9 (9) | 3 (4)
Leptospirosis (Infections and infestations) | 0 (0) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Lymphadenitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Measles (Infections and infestations) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis Aseptic (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Mumps (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Oral Herpes (Infections and infestations) | 2 (2) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis Media (Infections and infestations) | 2 (2) | 0 (0)
Otitis Media Chronic (Infections and infestations) | 0 (0) | 1 (1)
Paratyphoid Fever (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 32 (35) | 19 (25)
Pharyngitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 15 (15) | 4 (4)
Plasmodium Falciparum Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 33 (37) | 12 (12)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Measles (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Primary Atypical (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia Viral (Infections and infestations) | 1 (1) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 5 (5) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 4 (4) | 3 (3)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Scarlet Fever (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 12 (12) | 4 (4)
Tonsillitis Bacterial (Infections and infestations) | 2 (2) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Tuberculous Pleurisy (Infections and infestations) | 0 (0) | 1 (1)
Typhoid Fever (Infections and infestations) | 15 (18) | 13 (13)
Typhus (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (11) | 5 (6)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 22 (23) | 14 (17)
Varicella (Infections and infestations) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 32 (35) | 29 (29)
Viral Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Viral Rash (Infections and infestations) | 0 (0) | 3 (3)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Vulval Abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Adverse Event Following Immunisation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Arthropod Bite (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ear Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrical Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Eyeball Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 15 (16) | 6 (6)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Forearm Fracture (Injury, poisoning and procedural complications) | 9 (9) | 4 (4)
Foreign Body (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Foreign Body In Eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Genital Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Humerus Fracture (Injury, poisoning and procedural complications) | 9 (9) | 2 (2)
Impacted Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple Injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Near Drowning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Open Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Poisoning Deliberate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Adhesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Road Traffic Accident (Injury, poisoning and procedural complications) | 71 (75) | 38 (39)
Scrotal Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake Bite (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sports Injury (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Calcium Deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture Malunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatic Fever (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Angiofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Neoplasm Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Soft Tissue Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bone Giant Cell Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Ear Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lip Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Soft Tissue Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute Disseminated Encephalomyelitis (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Venous Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Complex Partial Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 4 (4) | 2 (2)
Convulsions Local (Nervous system disorders) | 1 (1) | 0 (0)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 8 (9) | 4 (7)
Extrapyramidal Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 13 (23) | 7 (7)
Grand Mal Convulsion (Nervous system disorders) | 2 (3) | 0 (0)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Intercostal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Migraine Without Aura (Nervous system disorders) | 1 (1) | 0 (0)
Partial Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1)
Tonic Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Viith Nerve Paralysis (Nervous system disorders) | 3 (3) | 0 (0)
Abortion Complete (Pregnancy, puerperium and perinatal conditions) | 3 (4) | 0 (0)
Abortion Incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Abortion Spontaneous Incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion Threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Breech Presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Cephalo-Pelvic Disproportion (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
False Labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Foetal Distress Syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Postpartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2)
Puerperal Pyrexia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abnormal Behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosomatic Disease (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 2 (2) | 1 (2)
Somatoform Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 2 (2)
Calculus Ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis Acute (Renal and urinary disorders) | 3 (3) | 1 (1)
Nephrotic Syndrome (Renal and urinary disorders) | 2 (4) | 0 (0)
Neurogenic Bladder (Renal and urinary disorders) | 0 (0) | 1 (3)
Post Streptococcal Glomerulonephritis (Renal and urinary disorders) | 9 (9) | 3 (3)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Tubular Acidosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Acquired Phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Ovarian Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Cervical Erosion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 (19) | 9 (9)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Child Abuse (Social circumstances) | 0 (0) | 1 (1)
Physical Assault (Social circumstances) | 4 (4) | 1 (1)
Victim Of Child Abuse (Social circumstances) | 0 (0) | 1 (1)
Victim Of Crime (Social circumstances) | 1 (1) | 1 (1)
Victim Of Sexual Abuse (Social circumstances) | 1 (1) | 0 (0)
Abortion Induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm Ruptured (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=1334) | Placebo Group (N=663)
Asthenia (General disorders) | 378 (530) | 167 (244)
Injection Site Erythema (General disorders) | 107 (142) | 52 (71)
Injection Site Pain (General disorders) | 616 (994) | 275 (449)
Injection Site Swelling (General disorders) | 68 (84) | 33 (36)
Malaise (General disorders) | 476 (689) | 239 (352)
Pyrexia (General disorders) | 267 (291) | 125 (137)
Nasopharyngitis (Infections and infestations) | 85 (113) | 45 (61)
Upper Respiratory Tract Infection (Infections and infestations) | 95 (104) | 54 (62)
Myalgia (Musculoskeletal and connective tissue disorders) | 414 (585) | 197 (296)
Headache (Nervous system disorders) | 567 (866) | 264 (409)
Cough (Respiratory, thoracic and mediastinal disorders) | 63 (69) | 48 (61)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 46 (48) | 36 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.